CLINICAL TRIAL: NCT00279188
Title: Asthma Management Project University Leiden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: The Netherlands Asthma Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AF 3.2.92.45, AMPUL; AF 3.2.92.45
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-01-19 (Estimated); Status verified 2004-09

CONDITIONS: Asthma
Keywords: Bronchial hyperresponsiveness; Atopy; Inhaled steroids; Exacerbations; Lung function decline; Prognosis
MeSH Terms: conditions — Asthma; Bronchial Hyperreactivity

INTERVENTIONS:
Procedure: Guiding therapy by bronchial hyperrsponsiveness

SUMMARY:
The long-term course of asthma shows variable outcome with regard to the incidence of exacerbations and the decline of lung function over time. The present study aimed:

1. to investigate whether asthma management additionally guided by the degree of bronchial hyperresponsiveness leads to a better outcome
2. to examine the predictors among clinical and inflammatory disease markers of the long-term decline in lung function

DETAILED DESCRIPTION:
Asthma is associated with a specific inflamma¬tory state of the airways. Assuming that the degree of airway inflammation is a determinant for the long-term disease outcome, it follows that, asthma therapy should be aimed at maximal reduction of airway inflammation, in addition to reducing symptoms. However, according to current guidelines, therapy should only be directed to the clinical severity of the disease. There is increasing evidence that bronchial hyper¬respon¬siveness can be used as a non-invasive reflection of airway inflamma¬tion [29]. However, it is still unknown whether bronchial responsiveness provides relevant additional information for adjusting therapy during follow-up of patients with asthma. Therefore, in this study we will:

1. compare the disease outcome in two parallel groups of patients with asthma, receiving therapy aimed at either clinical severity only, or therapy aimed at both clinical severity, and bronchial hyper¬responsiveness to methacho¬li¬ne. The outcome will be assessed at three levels. First, the severity, second, lung function and bronchial responsive¬ness, and third, humoral, cellular, and histological indices of airway inflamma¬tion. To that end we will assess symptoms, lung function, bronchial respon¬siveness, and immunological parameters in blood, every three months. Furthermore, a bronchos¬copy with a bronchoalveolar lavage and bronchial biopsy will be carried out to provide for material for immunologic and pathologic anatomical examination, at the beginning and at the end of the study.
2. analyse the predictors among clinical- and inflammatory parameters of exacerbations and long-term decline in lung function during long-term follow-up

ELIGIBILITY:
Inclusion Criteria:

* Asthma based on GINA guidelines (www.ginasthma.org)

Exclusion Criteria:

* oral steroids

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75
Dates: Start 1992-05; Study Completion 2008-09

PRIMARY OUTCOMES:
Exacerbations
Post-bronchodilator FEV1

SECONDARY OUTCOMES:
Bronchial hyperrsponsiveness
Airway inflammationn in bronchial biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Sterk, MD, PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Background] van Rensen EL, Sont JK, Evertse CE, Willems LN, Mauad T, Hiemstra PS, Sterk PJ; AMPUL Study Group. Bronchial CD8 cell infiltrate and lung function decline in asthma. Am J Respir Crit Care Med. 2005 Oct 1;172(7):837-41. doi: 10.1164/rccm.200504-619OC. Epub 2005 Aug 4. PMID 16085937
- [Background] Sont JK, Willems LN, Bel EH, van Krieken JH, Vandenbroucke JP, Sterk PJ. Clinical control and histopathologic outcome of asthma when using airway hyperresponsiveness as an additional guide to long-term treatment. The AMPUL Study Group. Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 1):1043-51. doi: 10.1164/ajrccm.159.4.9806052. PMID 10194144
- See also: Leiden University Medical Center — http://www.lumc.nl